CLINICAL TRIAL: NCT03770624
Title: An Open-Label Phase 1b Study to Evaluate the Dose-Related Safety, Efficacy, and Pharmacokinetic Profile of Different Doses of QL-007 in Chronic Hepatitis B Patients
Brief Title: A Study to Investigate the Safety, Efficacy and PK of Multiple Doses of QL-007 in Chronic Hepatitis B Patients in CHINA
Acronym: QL-007
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QL-007-003
Record Dates: First submitted 2018-06-20; First posted 2018-12-10 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-06

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 200 mg QD (Experimental): Tablet QL-007 will be administered orally daily (200 mg QD) over the 28 days under fasted state. Patients fast for 10h before administration and 1h after administration.
  Interventions: Drug: QL-007 tablet
- 400 mg QD (Experimental): Tablet QL-007 will be administered orally daily (400 mg QD) over the 28 days under fasted state. Patients fast for 10h before administration and 1h after administration.
  Interventions: Drug: QL-007 tablet
- 600 mg QD (Experimental): Tablet QL-007 will be administered orally daily (600 mg QD) over the 28 days under fasted state. Patients fast for 10h before administration and 1h after administration.
  Interventions: Drug: QL-007 tablet
- 100 mg BID (Experimental): Tablet QL-007 will be administered orally daily (100 mg BID) over the 28 days under fasted state. Patients fast for 2h before administration and 1h after administration.
  Interventions: Drug: QL-007 tablet
- 200 mg BID (Experimental): Tablet QL-007 will be administered orally daily (200 mg BID) over the 28 days under fasted state. Patients fast for 2h before administration and 1h after administration.
  Interventions: Drug: QL-007 tablet
- TDF 300 mg QD (Active Comparator): TDF will be administered orally daily (300 mg QD) over the 28 days not request fast .
  Interventions: Drug: TDF

INTERVENTIONS:
Drug: QL-007 tablet — QL-007 will be administered orally daily over the 28 days under fasted state.
  Arms: 100 mg BID; 200 mg BID; 200 mg QD; 400 mg QD; 600 mg QD
Drug: TDF — TDF will be administered orally daily over the 28 days e.
  Arms: TDF 300 mg QD

SUMMARY:
This is a randomized, open-label, positive-control, dose-escalation Phase 1b trial in 60 patients with chronic HBV infection to determine the safety, preliminary efficacy, and pharmacokinetics (PK) of QL-007 after administration over 28 days of multiple oral doses in a fasted state at the following planned dose levels: 200, 400, and then 600 mg.

DETAILED DESCRIPTION:
This is a randomized, open-label, positive-control, dose-escalation Phase 1b trial in 60 patients with chronic HBV infection to determine the safety, preliminary efficacy, and pharmacokinetics (PK) of QL-007 after administration over 28 days of multiple oral doses in a fasted state at the following planned dose levels: 200, 400, and then 600 mg.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Hepatitis B infection, defined as positive test for Hepatitis B surface antigen (HBsAg) for more than 6 months prior to randomization
* HBV DNA at screening greater than or equal to (>/=) 2 × 10^4 international units per milliliter (IU/mL) for Hepatitis B e antigen (HBeAg) positive participants, or >/=2 × 10^3 IU/mL for HBeAg-negative participants
* ALT> 1 x upper limit of normal (ULN) and < 10 x upper limit of normal (ULN)
* Anti-HBV treatment-naive adults; adults who have taken oral anti-HBV nucleoside therapy with the last dose ≥4 weeks prior to screening are also eligible.
* Signed informed consent.

Exclusion Criteria:

* Known co-infection with HIV, hepatitis C virus (HCV) or hepatitis D virus (HDV)
* Presence of autoimmune disorders
* History of liver disease other than Hepatitis B
* History of Gilbert's Disease
* Any sign of decompensated liver disease
* Known or suspected cirrhosis
* Evidence of hepatocellular carcinoma
* Patient has clinically significant, uncontrolled heart disease and/or recent cardiac event (within 6 months)
* Pregnant or lactating females
* Diabetes
* Alcohol or substance abuse
* History of bleeding diathesis
* Patients with a history of seizures, central nervous system disorders or psychiatric disability thought to be clinically significant in the opinion of the investigator.
* History of clinically significant gastrointestinal, cardiovascular, endocrine, renal, ocular, pulmonary, psychiatric or neurological disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-03-30 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in serum HBV DNA from baseline at Day3, 8, 15, 22 and 28 | Time Frame: Day 1, Day 3, Day 8, Day 15, Day 22 and Day 28
  Blood samples will be collected on Day -1 , 1, 3, 8, 15, 22, 28 and the follow-up 7 ±1 days

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of QL-007 following multiple doses | Days 1, 3, 8, 15, 22, and 28. On Days 1, 3, 8, 15, 22, and 28, samples will be collected predose; on Days 1 and 28, samples will also be collected at 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h and 24h postdose
  Concentrations of QL-007 in plasma will be collected on Day 1, Day 3, Day 8, Day 15, Day 22 and Day 28.
The time to Cmax (tmax) of QL-007 following multiple doses | Days 1, 3, 8, 15, 22, and 28. On Days 1, 3, 8, 15, 22, and 28, samples will be collected predose; on Days 1 and 28, samples will also be collected at 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h and 24h postdose
  Concentrations of QL-007 in plasma will be collected on Day 1, Day 3, Day 8, Day 15, Day 22 and Day 28.
AUC0-t (area under the plasma concentration versus time curve) of QL-007 following multiple doses | Days 1, 3, 8, 15, 22, and 28. On Days 1, 3, 8, 15, 22, and 28, samples will be collected predose; on Days 1 and 28, samples will also be collected at 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h and 24h postdose
  Concentrations of QL-007 in plasma will be collected on Day 1, Day 3, Day 8, Day 15, Day 22 and Day 28.
AUC0-∞ of QL-007 following multiple doses following multiple doses | Days 1, 3, 8, 15, 22, and 28. On Days 1, 3, 8, 15, 22, and 28, samples will be collected predose; on Days 1 and 28, samples will also be collected at 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h and 24h postdose
  Concentrations of QL-007 in plasma will be collected on Day 1, Day 3, Day 8, Day 15, Day 22 and Day 28.
t1/2 (terminal elimination half-life) of QL-007 following multiple doses | Days 1, 3, 8, 15, 22, and 28. On Days 1, 3, 8, 15, 22, and 28, samples will be collected predose; on Days 1 and 28, samples will also be collected at 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h and 24h postdose
  Concentrations of QL-007 in plasma will be collected on Day 1, Day 3, Day 8, Day 15, Day 22 and Day 28.
Vz/F(apparent volume of distribution for the terminal disposition phase) of QL-007 following multiple doses | Days 1, 3, 8, 15, 22, and 28. On Days 1, 3, 8, 15, 22, and 28, samples will be collected predose; on Days 1 and 28, samples will also be collected at 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h and 24h postdose
  Concentrations of QL-007 in plasma will be collected on Day 1, Day 3, Day 8, Day 15, Day 22 and Day 28.
Change in serum HBsAg from baseline at Day 1, Day 3, Day 8, Day 15, Day 22 and Day 28 | Time Frame: Day 1, Day 3, Day 8, Day 15, Day 22 and Day 28
  Blood samples will be collected on Day -1 , 1, 3, 8, 15, 22, 28 and the follow-up 7 ±1 days
adverse events (AEs) | From randomization up to Day 35
  AEs occur during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No